CLINICAL TRIAL: NCT05731843
Title: A Phase 1, Open-Label Study to Evaluate the Potential Drug-Drug Interaction Between Bemnifosbuvir and Ruzasvir and Food-Drug Interaction in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Ruzasvir and Bemnifosbuvir
Acronym: AT-527
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-003
Record Dates: First submitted 2023-02-09; First posted 2023-02-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — ruzasvir; AT-511

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BEM vs BEM + Ruzasvir n=16 (Experimental)
  Interventions: Drug: Cohort 1 BEM + Ruzasvir
- Ruzasvir vs Ruzasvir + BEM n=16 (Experimental)
  Interventions: Drug: Cohort 2 Ruzasvir + BEM

INTERVENTIONS:
Drug: Cohort 1 BEM + Ruzasvir — Days 1 to 6 BEM under fasting conditions. Days 7 to 12 of BEM and Ruzasvir coadministered under fasting conditions. Days 13 to 18 of BEM and Ruzasvir coadministered under fed conditions
  Other Names: AT-527
  Arms: BEM vs BEM + Ruzasvir n=16
Drug: Cohort 2 Ruzasvir + BEM — Days 1 to 6 of Ruzasvir under fasting conditions. Days 7 to 12 of Ruzasvir and BEM coadministered under fasting conditions. Days 13 to 18 of Ruzasvir and BEM coadministered under fed conditions
  Other Names: AT-527
  Arms: Ruzasvir vs Ruzasvir + BEM n=16

SUMMARY:
Drug-drug interaction study of Ruzasvir and Bemnifosbuvir

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug.
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days of dosing.
* Concomitant use of prescription medications, or systemic over-the-counter medications.
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of BEM | Days 6, 12, 18
  Maximum plasma concentration (Cmax) and Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of Ruzasvir | Days 6, 12, 18
  Maximum plasma concentration (Cmax) and Area under the plasma concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Quebec, Canada